CLINICAL TRIAL: NCT03693742
Title: Evaluation of Monosodium Glutamate (MSG) to Reduce Salivary Gland and Renal Accumulation of PSMA-binding Radiopharmaceuticals
Brief Title: MSG Use With 18F-DCFPyL PET/CT Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: H18-02227
Record Dates: First submitted 2018-09-27; First posted 2018-10-03 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2021-11

CONDITIONS: Prostate Cancer; Prostate Cancer Metastatic; Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective double blind intra-participant comparison of [18F]-DCFPyL PET/CT scans performed after orally administered MSG or placebo. The participants will receive oral administration of MSG or placebo, in two different examination sessions, 30 minutes before [18F]-DCFPyL injection.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: For randomization, a computer generated random list will determine the order of the scans (MSG first, placebo first). Sealed envelopes will be prepared. A study coordinator or technologist not involved in measuring vital signs or collecting adverse events will prepare the tomato juice solution based on the randomization envelope. The rest of the team will not be informed of which tomato juice is used (placebo or MSG) but this information will be recorded and will be immediately accessible should a participant experience a severe adverse event.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18F-DCFPyL PET/CT scan with MSG drink (Experimental): Food grade MSG will be dissolved in low sodium tomato juice, and administered orally before 18F-DCFPyL administration.
  Interventions: Diagnostic Test: 18F-DCFPyL PET/CT scan; Other: MSG drink
- 18F-DCFPyL PET/CT scan with placebo drink (Placebo Comparator): Regular tomato juice will be used, and administered orally before 18F-DCFPyL administration.
  Interventions: Diagnostic Test: 18F-DCFPyL PET/CT scan; Other: Placebo drink

INTERVENTIONS:
Diagnostic Test: 18F-DCFPyL PET/CT scan — Participants will have their weight recorded and baseline vital signs (blood pressure, heart rate, and oxygen saturation level) measured prior to the tomato juice ingestion, immediately prior to 18F-DCFPyL injection and 5 to 15 minutes after injection.
  The participant will receive a bolus intravenous dose of 18F-DCFPyL.
  After 60 min, the vital signs will be recorded and again two hours after 18F-DCFPyL. Immediately before scanning, the participants will be taken to a designated washroom and asked to void.
  The PET/CT image acquisition time will be approximately 30 minutes.
Other: Placebo drink — Participants will consume 300mL of tomato juice 30 minutes prior to 18F-DCFPyL injection.
  Arms: 18F-DCFPyL PET/CT scan with placebo drink
Other: MSG drink — Participants will consume 300mL of tomato juice with MSG 30 minutes prior to 18F-DCFPyL injection.
  Arms: 18F-DCFPyL PET/CT scan with MSG drink

SUMMARY:
18F-DCFPyL is an agent that binds to prostate specific membrane antigen (PSMA). Due to high levels of PSMA in prostate cancer, treatments targeting PSMA have been developed to deliver therapy to these specific target cells. Unfortunately when this treatment is delivered there is radiotracer uptake in the salivary glands and kidneys, not related to cancer, which causes dry mouth and causes patients to stop treatment. It is proposed that having tomato juice containing monosodium glutamate (MSG) may reduce radiotracer uptake in the salivary glands and kidneys and reduce damage to these tissues.

DETAILED DESCRIPTION:
This is a prospective single cohort study to evaluate the utility of MSG in reducing salivary gland radiotracer uptake, in patients who undergo an 18F-DCFPyL Positron Emission tomography / Computer Tomography (PET/CT) scan.

18F-DCFPyL PET/CT scans Each participant will receive 2 18F-DCFPyL PET/CT scans at the BC Cancer - Vancouver Centre, as part of this research sub-study. Each participant will receive tomato juice before each appointment. One visit they will have tomato juice containing MSG and the other will be a placebo (standard tomato juice).

Each study participant will receive a bolus intravenous dose of 18F-DCFPyL. The participant will rest in a comfortable chair for 120 minutes and will then be taken to the PET/CT scanner for images.

24 hour follow-up All participants will be requested to either return to the functional imaging department approximately 24 hours (acceptable range 16-28 hours) after the injection of 18F-DCFPyL and tomato juice consumption or agree to be contacted by phone. The participants will be asked if they experienced any undesirable effects following the administration of 18F-DCFPyL and tomato juice, or in the intervening 24 hours. The local site attending nuclear medicine physician will then make an assessment as to whether these effects are likely related to 18F-DCFPyL and/or tomato juice administration.

The study is expected to take approximately 1 year for accrual.

ELIGIBILITY:
Inclusion Criteria:

* Known prostate cancer with biochemical recurrence after initial curative therapy with radical prostatectomy, presenting with a prostate specific antigen (PSA) greater than 0.4 ng/mL.
* Subjects with findings on other examinations (such as plain x-ray, CT, MRI or bone scintigraphy and others) that are suspicious for metastatic disease but not conclusively diagnostic of metastatic disease, within 3 months of PET scan.
* Known prostate cancer with biochemical recurrence after initial curative therapy with radiation therapy (including brachytherapy), with a PSA level >2 ng/mL above the nadir after radiation therapy.
* Castration resistant prostate cancer with a minimum PSA of 2.0 ng/mL with 2 consecutive rises above the nadir and castrate levels of testosterone (<1.7 nmol/L). Treatment does not need to be discontinued before the 18F-DCFPyL scan.
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less.

Exclusion Criteria:

* Medically unstable (eg. acute illness, unstable vital signs)
* Unable to lie supine for the duration of imaging
* Unable to provide written consent
* Exceeds safe weight limit of the PET/CT bed (204.5 kg) or unable to fit through the PET/CT bore (diameter 70 cm)
* Severe uncontrolled hypertension (systolic blood pressure above 140 mm Hg and diastolic blood pressure above 90 mm Hg, or systolic blood pressure above 180 mm Hg, or diastolic blood pressure above 110 mg Hg). Patients with controlled hypertension under medication are eligible
* History of severe asthma that has led to hospitalizations or emergency room visits
* History of intolerance to MSG
* History of severe headaches or migraines triggered by food or MSG
* Participants on a sodium/salt restricted diet due to other medical conditions
* No new treatment has started between the first and second 18F-DCFPyL PET/CT

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois Benard, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The effects of monosodium glutamate on PSMA radiotracer uptake in men with recurrent prostate cancer: a prospective, randomized, double-blind, placebo-controlled intra-individual imaging study. — http://jnm.snmjournals.org/content/early/2020/05/07/jnumed.120.246983.abstract

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Biochemically recurrent prostate cancer patients were screened from a PSMA study wait list, for eligibility between November 1, 2019 and December 1, 2019 at BC Cancer, Vancouver BC. 10 participants were enrolled between November 4th 2019, and December 5th 2019.
Pre-assignment Details: 10 of 10 participants were randomized.
Groups:
- MSG, Then Placebo: After a fasting period of 4 hours, participants first received oral administration of 12.7 g of food grade MSG dissolved in 300 mL low sodium tomato juice, prior to receiving the 18F-DCFPyL radio-tracer administration for their PET/CT scan.
  Within 1 week, participants returned and after having fasted for 4 hours, then received oral administration of the Placebo (300 mL regular sodium tomato juice) prior to receiving the 18F-DCFPyL radio-tracer administration for their PET/CT scan.
- Placebo, Then MSG: After a fasting period of 4 hours, participants first received oral administration of the Placebo (300 mL regular sodium tomato juice) prior to receiving the 18F-DCFPyL radio-tracer administration for their PET/CT scan.
  Within 1 week, participants returned and after having fasted for 4 hours, then received oral administration of 12.7 g of food grade MSG dissolved in 300 mL low sodium tomato juice, prior to receiving the 18F-DCFPyL radio-tracer administration for their PET/CT scan.
Period: Overall Study
Arm/Group | MSG, Then Placebo | Placebo, Then MSG
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MSG, Then Placebo | Placebo, Then MSG | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 7 | 3 | 10
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 7 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Salivary Gland Maximal Standardized Uptake Values Corrected for Lean Body Mass (SULmax) for 18F-DCFPyL
Description: Comparison of MSG and placebo 18F-DCFPyL salivary gland (submandibular) accumulation measured by the maximal standardized uptake values corrected for lean body mass (SULmax). For determination of salivary gland uptake, regions of interest will be drawn around the salivary glands, using a standardized contouring method, to measure the SULmax. The average SULmax in the organs will be used for this analysis.
Time Frame: scan with MSG and 3-7 days later, scan with Placebo (or vice versa)
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the efficacy analysis.
Measure: Mean (Standard Deviation); unit: SULmax
Groups:
- 18F-DCFPyL PET/CT Scan With MSG Drink: Participants who received MSG dissolved in juice, in a fasting state, prior to the administration of 18F-DCFPyL, in either the first or second PET/CT scan.
- 18F-DCFPyL PET/CT Scan With Placebo Drink: Participants who received the Placebo juice, in a fasting state, prior to the administration of 18F-DCFPyL, in either the first or second PET/CT scan.
Arm/Group | 18F-DCFPyL PET/CT Scan With MSG Drink | 18F-DCFPyL PET/CT Scan With Placebo Drink
Number analyzed (Participants) | 10 | 10
SULmax | 9.9 (4.8) | 15.1 (6.2)
Statistical Analysis 1: Comparison: 18F-DCFPyL PET/CT Scan With MSG Drink vs 18F-DCFPyL PET/CT Scan With Placebo Drink; Null hypothesis is that there was no difference in uptake of F18-DCFPyL between the MSG and placebo groups. A sample size of 10 achieves 100% power to detect a mean of paired differences of 5.0 (33%) with an estimated standard deviation of differences of 1.0 and with a significance level (alpha) of 0.05 using a one-sided paired t-test. If the estimated standard deviation of differences is 5.0, a sample size of 10 achieves 90% power to detect a mean difference of 5.0 with an alpha of 0.05; Test type: Superiority; p < 0.001, Mixed Models Analysis — A P value of less than 0.05 was considered significant

2. Secondary Outcome: Renal Maximal Standardized Uptake Values Corrected for Lean Body Mass (SULmax) for 18F-DCFPyL
Description: Comparison of MSG and placebo 18F-DCFPyL renal accumulation measured by the maximal standardized uptake values corrected for lean body mass (SULmax). For determination of renal uptake, regions of interest will be drawn around the kidneys, using a standardized contouring method, to measure the SULmax. The average SULmax in the organs will be used for this analysis.
Time Frame: scan with MSG and 3-7 days later, scan with Placebo (or vice versa)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SULmax
Arm/Group | 18F-DCFPyL PET/CT Scan With MSG Drink | 18F-DCFPyL PET/CT Scan With Placebo Drink
Number analyzed (Participants) | 10 | 10
SULmax | 27.4 (8.0) | 37.5 (9.6)

3. Secondary Outcome: Tumour Maximal Standardized Uptake Values Corrected for Lean Body Mass (SULmax) for 18F-DCFPyL
Description: Comparison of MSG and placebo 18F-DCFPyL tumour accumulation measured by the maximal standardized uptake values corrected for lean body mass (SULmax). For determination of tumour uptake, all malignant lesions, the SULmax were measured using the PET Edge tool running on MIM. All regions of interest were created in one dataset by a blinded observer, and then saved and compared to the identical location in the second dataset for matched comparisons of activity. The median SULmax in the malignant lesions will be used for this analysis.
Time Frame: scan with MSG and 3-7 days later, scan with Placebo (or vice versa)
Population: as for outcome 1
Measure: Median (Full Range); unit: SULmax
Units Other Than Participants: malignant lesions
Arm/Group | 18F-DCFPyL PET/CT Scan With MSG Drink | 18F-DCFPyL PET/CT Scan With Placebo Drink
Number analyzed (Participants) | 10 | 10
Number analyzed (malignant lesions) | 140 | 142
SULmax | 2.8 [0.7 to 23.4] | 4.4 [1.1 to 30.3]

4. Secondary Outcome: Number of Participants With Tomato Juice (Containing Either MSG or Placebo) Related Adverse Events as Assessed by Abnormal Vital Sign Measurement.
Description: Vital signs (blood pressure, heart rate and pulse oximetry) will be measured at two time points (before tomato juice and 2 hours after radiotracer injection). All values that fall outside of the normal parameters will be assessed by a physician and reported as an adverse event.
Time Frame: 2 hours
Measure: Count of Participants; unit: Participants
Groups:
- MSG Intervention: After a fasting period of 4 hours, participants first received oral administration of 12.7 g of food grade MSG dissolved in 300 mL low sodium tomato juice, prior to receiving the 18F-DCFPyL radio-tracer administration for their PET/CT scan.
- Placebo Intervention: After a fasting period of 4 hours, participants first received oral administration of the Placebo (300 mL regular sodium tomato juice) prior to receiving the 18F-DCFPyL radio-tracer administration for their PET/CT scan.
Arm/Group | MSG Intervention | Placebo Intervention
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- 18F-DCFPyL PET/CT Scan With MSG Drink: Food grade MSG will be dissolved in low sodium tomato juice, and administered orally before 18F-DCFPyL administration.
  18F-DCFPyL PET/CT scan: Participants will have their weight recorded and baseline vital signs (blood pressure, heart rate, and oxygen saturation level) measured prior to the tomato juice ingestion, immediately prior to 18F-DCFPyL injection and 5 to 15 minutes after injection.
  The participant will receive a bolus intravenous dose of 18F-DCFPyL.
  After 60 min, the vital signs will be recorded and again two hours after 18F-DCFPyL. Immediately before scanning, the participants will be taken to a designated washroom and asked to void.
  The PET/CT image acquisition time will be approximately 30 minutes.
  MSG drink: Participants will consume 300mL of tomato juice with MSG 30 minutes prior to 18F-DCFPyL injection.
- 18F-DCFPyL PET/CT Scan With Placebo Drink: Regular tomato juice will be used, and administered orally before 18F-DCFPyL administration.
  18F-DCFPyL PET/CT scan: Participants will have their weight recorded and baseline vital signs (blood pressure, heart rate, and oxygen saturation level) measured prior to the tomato juice ingestion, immediately prior to 18F-DCFPyL injection and 5 to 15 minutes after injection.
  The participant will receive a bolus intravenous dose of 18F-DCFPyL.
  After 60 min, the vital signs will be recorded and again two hours after 18F-DCFPyL. Immediately before scanning, the participants will be taken to a designated washroom and asked to void.
  The PET/CT image acquisition time will be approximately 30 minutes.
  Placebo drink: Participants will consume 300mL of tomato juice 30 minutes prior to 18F-DCFPyL injection.
Arm/Group | 18F-DCFPyL PET/CT Scan With MSG Drink | 18F-DCFPyL PET/CT Scan With Placebo Drink
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT03693742/Prot_SAP_000.pdf